CLINICAL TRIAL: NCT06166238
Title: Comparative Study Between Millard and Tennison Randall Techniques in Complete and Incomplete Cleft Lip Repair.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif Abdelnaser Ibrahim, Resident doctor at Plastic & Reconstructive surgery at Assiut university, Assiut University
Other Study IDs: Unilater cleft lip.
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cleft Lip, Unilateral
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Patients who will be subjected to Millard Technique
  Interventions: Procedure: Millard and Tension Randal Technique
- Group II: patients who will be subjected to Tension Randal
  Interventions: Procedure: Millard and Tension Randal Technique

INTERVENTIONS:
Procedure: Millard and Tension Randal Technique — Millard recognized that the majority of Cupid's bow, one philtral column, and the philtral dimple were intact on the medial aspect of a unilateral cleft lip but required rotation to shift the tissue into a normal anatomic position (Millard, 1964b) The Tennison-Randall technique involves a back-cut that extends from the cleft Cupid's bow peak toward the center of the philtrum that is filled by a laterally based triangular flap whose width is the measured deficiency in lip height.

SUMMARY:
"the investigators will compare the quantitative and qualitative (functional and aesthetic outcomes) of these two surgical approaches for repair of the unilateral cleft lip using an evaluation protocol developed many years ago by the research council of Operation Smile, a non- profit organization based in Virginia Beach, USA. Operation Smile delivers charity management of cleft lip and palate cases in many different developing countries around the world. Under this protocol, a dual rating system has been developed with two scores: one preoperative score concerning the severity of cleft and one score for the postoperative results.

DETAILED DESCRIPTION:
One of the common congenital malformations in the head and neck is cleft lips. The prevalence of cleft lip is about 1:1000 of live birth; it also more common in boys and tends to present on the left side with a 6:3:1 ratio of left to right to bilateral. Many facial malformations, including cleft lip, are linked with environmental, maternal, and genetic factors, such as exposure to teratogen drugs, including isotretinoin, alcohol, or anticonvulsants. Similarly, some habits or diseases during pregnancy increase the risk of the cleft lip as smoking, pregestational and gestational diabetes, and specific nutritional deficiencies. The treatment begins soon after the child's birth and continues until adulthood. The purpose of cleft treatment is aesthetic and functional rehabilitation. Surgical repair is important for facial growth preservation, normal speech formation and development of proper dentition. The less number of interventions, the less the scaring results and hence, growth retardation Nowadays, the most commonly used techniques in managing unilateral cleft lip (UCL) are Millard's rotation advancement and Tennison Randall's triangular flap repairs. This study aimed to use anthropometric analysis by anthropometric measurements taken pre and post operation to evaluate the quantitative assessment of the modified Millard technique compared with the Tennison Randall technique in UCL repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients are generally fit
* Patients with unilateral with or without cleft palate
* Patients with compliance for follow up.

Exclusion Criteria:

* Syndromic cases.
* Patients are generally unfit.
* Secondary cleft lip.
* Age less than 3 months, more than 4 years
* Bilateral cleft lip.

Ages: 3 Months to 6 Months | Sex: All
Age Groups: Child
Study Population: Patients with complete and incomplete unilateral cleft lip.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
functional and aesthetic outcomes after repair | 6 months
  two scores: one preoperative score concerning the severity of cleft and one score for the Assessment of the results based on the post-operative scoring sheet included items for evaluating the integrity and symmetry of the Cupid's bow, nasal symmetry, lateral lip symmetry, vermilion contour, and white roll continuity. The individual scores for each factor were combined to yield an overall rating of poor, fair, good, and excellent.

REFERENCES:
- [Background] Willhite CC, Hill RM, Irving DW. Isotretinoin-induced craniofacial malformations in humans and hamsters. J Craniofac Genet Dev Biol Suppl. 1986;2:193-209. PMID 3491113
- [Result] Parker SE, Mai CT, Strickland MJ, Olney RS, Rickard R, Marengo L, Wang Y, Hashmi SS, Meyer RE; National Birth Defects Prevention Network. Multistate study of the epidemiology of clubfoot. Birth Defects Res A Clin Mol Teratol. 2009 Nov;85(11):897-904. doi: 10.1002/bdra.20625. PMID 19697433
- [Result] Jones MC. Facial clefting. Etiology and developmental pathogenesis. Clin Plast Surg. 1993 Oct;20(4):599-606. PMID 8275626